CLINICAL TRIAL: NCT00820768
Title: A Phase I of ABI-010 (Nab-17-AAG) and ABI-007 (Abraxane) Administered Weekly in Patients With Advanced Non-Hematologic Malignancies
Brief Title: A Trial of ABI-010 & ABI-007 in Patients With Advanced Non-Hematologic Malignancies
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA501
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Solid Tumor
MeSH Terms: interventions — tanespimycin; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABI-010 (Experimental)
  Interventions: Drug: ABI-010

INTERVENTIONS:
Drug: ABI-010 — 17-AAG and ABI-007
  Other Names: 17-AAG and ABI-007

SUMMARY:
To determine MTD and DLT of ABI-010 given weekly every three weeks followed by one week of rest (Cycle 1). Determine MLD and DLT in combination with ABI-007; to characterize the toxicities of ABI-010 alone and in combination with ABI-007.

ELIGIBILITY:
Inclusion Criteria: Each subject must meet the following criteria to be enrolled in this study:

1. Pathologically confirmed advanced solid tumor malignancy.
2. Measurable or evaluable advanced solid tumors.
3. Patients with advanced solid tumor malignancy who failed standard therapy or for whom no standard therapy exists. Patients failing standard therapy should have received no more than 3 prior chemotherapy regimens.
4. Patients must have recovered for at least 3 weeks from prior treatment regimens and have no residual toxicity > Grade 2 (with the exception of peripheral neuropathy which must have improved to ≤ Grade 1).
5. Patient should have full recovery from any reversible side effects of prior chemotherapy.
6. Patient should have full recovery for at least 4 weeks since major surgery.
7. ECOG performance status 0-2.
8. Age ≥18 years.
9. Patient must have the following blood counts at Baseline:

   * WBC ≥ 3.0 x 10 cells/L.
   * ANC ≥ 1.5 x 10 cells/L.
   * Platelets ≥ 100 x 10 cells/L.
   * Hgb ≥ 9grams/dL.
10. Patient must have the following blood chemistry levels at Baseline:

    * AST (SGOT), ALT (SGPT) ≤ 1.5x upper limit of normal range (ULN);
    * Total Bilirubin ≤ ULN;
    * Alkaline phosphatase ≤ 2.5x ULN (unless bone metastasis is present in the absence of liver metastasis;
    * Creatinine ≤ 1.5 mg/dL
11. Peripheral neuropathy Grade ≤ 1 by NCI CTCAE V3.0.
12. Female of childbearing potential with negative serum pregnancy test within 72 hours prior to the first dose of study drug.
13. Males and females with reproductive potential must agree to utilize contraception considered adequate and appropriate by the investigator (including one barrier method) for the duration of the study and for 2 months after the end of study.
14. Life expectancy ≥ 3 months.
15. Informed consent document has been obtained.
16. If obese, a patient must be treated with doses calculated using his/her actual BSA (the physician must be comfortable treating at the full BSA dose regardless of BSA).

Exclusion Criteria: Subjects who meet any of the following criteria will be excluded from the study.

1. Concurrent therapy (chemotherapy, hormonal therapy, kinase inhibitors, immunotherapy, etc) for advanced solid tumor.
2. Patients receiving known CYP450 3A4 inhibitors.
3. Bisphosphonate therapy is allowed, however, patients should be stable on their current bisphosphonate, with no change, start or stop of treatment within 4 weeks prior to enrollment.
4. Patients with known brain metastases or leptomeningeal tumor involvement should be excluded from this clinical trial.
5. Uncontrolled intercurrent illness including, but not limited to, serious ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/ social situations that would limit compliance with study.
6. Patients with significant cardiovascular disease including congestive heart failure (New York Heart Association Class III or IV), active angina pectoris or recent myocardial infarction (within the last 6 months).
7. History of other malignancy within the last 5 years which would affect the diagnosis or assessment of advanced solid tumor excluding non-melanomatous skin cancer and cervical carcinoma.
8. Patients who have received an investigational drug within the previous 3 weeks.
9. Patient is currently enrolled in any other clinical study in which investigational procedures are performed or investigational therapies are administered. A patient may not enroll in such clinical trials while participating in this study.
10. Pregnant or nursing women.
11. Patients with history of allergy or hypersensitivity to the study drug or its excipients.
12. Patients with marked baseline prolongation of QT/QTc interval (>450 milliseconds).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2013-04-01 (Estimated); Study Completion 2014-04-01 (Estimated)

PRIMARY OUTCOMES:
The primary objectives of this study are to determine the maximum tolerated dose (MTD) and dose-limiting toxicities (DLTs) of ABI-010 given weekly for 3 weeks followed by 1 week of rest (Cycle 1); to determine MTD and DLTs of ABI-010 given in combination | EOS and Follow-Up

SECONDARY OUTCOMES:
To determine the pharmacokinetic parameters for ABI-010 when given on a weekly schedule alone and in combination with ABI-007; determine preliminary efficacy of ABI-010 when given on a weekly schedule in combination with ABI-007 | EOS and Follow-Up

CONTACTS AND LOCATIONS:
Overall Officials: Henry C. Pitot, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States